CLINICAL TRIAL: NCT06027008
Title: Mechanical Insufflation-Exsufflation (Cough Assist) in Critically Ill Adults (ACACIA)-a Randomized Clinical Feasibility Trial
Brief Title: Mechanical Insufflation-Exsufflation (Cough Assist) in Critically Ill Adults
Acronym: ACACIA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low inclusion rate: 7 patients since October 2023. Strict exclusion criteria limited potential participants. Current machine is discontinued, the department will acquire a different cough machine, impacting training and materials.
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACACIA
Record Dates: First submitted 2023-02-06; First posted 2023-09-07 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Critically Ill
Keywords: Mechanical insufflation-exsufflation; Cough Assist
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Randomized feasibility trial
Masking Description: Due to the nature of the intervention, blinding of healthcare professionals and any research personnel involved in the delivery of the intervention is not possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical Insufflation-Exsufflation (Experimental): Invasively ventilated patients will receive MI-E until successful extubation or for a maximum of 7 days. MI-E will be given in the morning and afternoon each calendar day. Patients will be pre-oxygenated with FiO2 100% prior to disconnection from the ventilator; additional 15 litres oxygen can be added; A pre-set program is used: three times three cycles with a 2-second insufflation and an immediate 2-second exsufflation. The cycles of the MI-E session will be performed with a positive and negative pressure of 40 cmH2O. The program is set up with the possibility of auto-triggering by the patient.
  Interventions: Device: Mechanical Insufflation-Exsufflation
- Standard airway care (No Intervention): Patients in the control group will receive usual airway care which includes endotracheal suctioning and manual hyperinflation used when indicated based on clinical signs as part of regular airway care. Care protocols for endotracheal suctioning and manual hyperinflation are predefined. As with the intervention arm, there will be no use of saline instillation during suctioning. Manual hyperinflation technique is described in the care protocol of the intensive care unit and ICU nurses are trained to perform this technique.

INTERVENTIONS:
Device: Mechanical Insufflation-Exsufflation — MI-E will be applied twice a day in invasively ventilated patients. Since the severity of illness can change in the ICU, each day the attending nurse will check for clinical reasons to not apply MI-E with regard to safety. The following clinical criteria are predefined as a reason to refrain from MI-E at that day:
  * severe ventilator instability (requiring > 12 cm H2O PEEP and dependency of > 60% FiO2);
  * severe hemodynamic instability (a need for large and sustained increase in continuous administration of intravenous vasopressive medication that are adjusted on a frequent basis in each nursing shift);
  * extra corporal membrane oxygenation (ECMO); and
  * deeply sedated patient (RASS score ≤ -4).
  Other Names: Cough assist
  Arms: Mechanical Insufflation-Exsufflation

SUMMARY:
The goal of this randomized feasibility trial is to evaluate the feasibility of Mechanical Insufflation-Exsufflation (MI-E) in invasively ventilated critically ill patients.

The main question[s] it aims to answer are:

* Is MI-E feasible?
* Is MI-E safe?

Participants in the intervention group will receive:

* MI-E
* Airway secretions will be removed by endotracheal suctioning, as part of routine airway care.
* Manual hyperinflation will only be used when necessary in an emergency situation. Patients in the control group will receive endotracheal suctioning and manual hyperinflation when clinically indicated.

The primary outcome is the proportion of delivered MI-E sessions (2 times per calendar day a MI-E session of 3 x 3 cycles of an in- and exsufflation) per patient according to study protocol (feasibility). Secondary outcomes are the total number of serious adverse events in relation to MI-E (safety) and preliminary exploratory data on the need for airway care interventions and clinical outcomes including duration of invasive ventilation, length of stay in ICU and mortality (efficacy).

DETAILED DESCRIPTION:
Bedside nurses, trained in using the MI-E device, will apply MI-E sessions at two moments per calendar day (morning and afternoon) for a maximum of 7 days while a patient is invasively ventilated.

MI-E settings are a 2-second insufflation and an immediate 2-second exsufflation. The cycles of the MI-E session will be performed with a positive and negative pressure of 40 cmH2O. The program is set up with the possibility of auto-triggering by the patient.

ELIGIBILITY:
Inclusion Criteria:

* admission to one of the participating ICUs;
* receiving invasive mechanical ventilation via an endotracheal tube; and
* expected to need invasive ventilation for more than 48 hours from consideration for inclusion.

Exclusion Criteria:

* use of MI-E before hospital admission, i.e., at home;
* known presence of bullous emphysema;
* known bronchopleural fistula;
* known pneumothorax or pneumomediastinum;
* known rib fractures;
* known barotrauma;
* known unstable spinal fractures;
* unsecured subarachnoidal haemorrhage;
* uncontrollable intracranial pressures; and
* any infection, or colonization with pathogens that requires strict aerogenic isolation. With an exception for patients in cohort isolation due to COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
intervention delivery | max. 7 days
  the proportion of complete sessions of MI-E every calender day (i.e. two MI-E sessions with 3 x 3 cycles of an in- and exsufflation) for all patients with a maximum of seven days of invasive ventilation

SECONDARY OUTCOMES:
incidence of pneumothorax (safety) | max 7 days
  incidence of pneumothorax for which drainage is needed attributed to MI-E or to routine airway care procedures (i.e., manual hyperinflation)
incidence of endotracheal tube obstruction (safety) | max 7 days
  incidence of endotracheal tube obstruction due to mucus plugging attributed to MI-E or regular airway care
incidence of severe hypoxemia (safety) | max 7 days
  incidence of severe hypoxemia
incidence of severe hypotension (safety) | max 7 days
  incidence of severe hypotension
incidence of severe hypertension (safety) | max 7 days
  incidence of severe hypertension
Acceptability of Intervention Measure (AIM) | through study completion, estimated one year
  1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Response scale 1 (completely disagree) - 5 (completely agree)
Intervention Appropriateness Measure (IAM) | through study completion, estimated one year
  1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Response scale 1 (completely disagree) - 5 (completely agree)
Feasibility of Intervention Measure (FIM) | through study completion, estimated one year
  1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Response scale 1 (completely disagree) - 5 (completely agree)
amount of time needed for MI-E (feasibility) | maximum of 1 hour per session
  time needed to deliver the MI-E intervention
endotracheal suctioning (feasibility) | max. 7 days
  frequency of endotracheal suctioning per ventilation day
MH (feasibility of MI-E) | max. 7 days
  frequency of manual hyperinflation
VAP (efficacy MI-E sample size calculation) | 28 days after inclusion
  incidence of ventilator associated pneumonia (VAP)
duration MV (efficacy MI-E sample size calculation) | 28 days after inclusion
  duration of invasive ventilation
Mortality day 28 (efficacy MI-E sample size calculation) | up to day 28 from ICU admission
  mortality at day 28
VFD-28 (efficacy MI-E sample size calculation) | 28 days after inclusion
  ventilator-free days at day 28
ICU mortality (efficacy MI-E sample size calculation) | 28 days after inclusion
  ICU mortality
hospital mortality (efficacy MI-E sample size calculation) | 28 days after inclusion
  hospital mortality
supplemental oxygen (efficacy MI-E sample size calculation) | 28 days after inclusion
  use of supplemental oxygen on ICU delivery after detubation
LOS ICU (efficacy MI-E sample size calculation) | 28 days after inclusion
  length of stay in ICU
LOS hospital (efficacy MI-E sample size calculation) | 28 days after inclusion
  length of stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Frederique Paulus, RN, PHD, Principal Investigator — Amsterdam UMC - intensive care
Locations (1):
- Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA), Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
Currently, there is no decision on a data sharing plan

REFERENCES:
- [Background] Stilma W, Verweij L, Spek B, Scholte Op Reimer WJM, Schultz MJ, Paulus F, Rose L. Mechanical insufflation-exsufflation for invasively ventilated critically ill patients-A focus group study. Nurs Crit Care. 2023 Nov;28(6):923-930. doi: 10.1111/nicc.12858. Epub 2022 Dec 4. PMID 36464804
- [Background] Swingwood EL, Stilma W, Tume LN, Cramp F, Voss S, Bewley J, Ntoumenopoulos G, Schultz MJ, Scholte Op Reimer W, Paulus F, Rose L. The Use of Mechanical Insufflation-Exsufflation in Invasively Ventilated Critically Ill Adults. Respir Care. 2022 Aug;67(8):1043-1057. doi: 10.4187/respcare.09704. Epub 2022 May 24. PMID 35610033
- [Background] Rose L, Adhikari NK, Leasa D, Fergusson DA, McKim D. Cough augmentation techniques for extubation or weaning critically ill patients from mechanical ventilation. Cochrane Database Syst Rev. 2017 Jan 11;1(1):CD011833. doi: 10.1002/14651858.CD011833.pub2. PMID 28075489